CLINICAL TRIAL: NCT06448689
Title: Prospective, Hybrid, Single-Center, Single-Arm Study to Characterize Sleep and Scratching Behavior in Adolescents and Adults With Atopic Dermatitis and Adults With Psoriasis
Brief Title: Analytical Validation of Wrist-Based Assessment of Nocturnal Scratch in Atopic Dermatitis and Psoriasis
Acronym: DECODE-Scratch
Status: Recruiting | Type: Observational
Sponsor: ActiGraph L.L.C (Industry)
Responsible Party: Sponsor
Other Study IDs: AG0001
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Atopic Dermatitis; Psoriasis
Keywords: nocturnal scratch; itch; validation; sleep impairment; pruritis
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis; Pruritus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pruritis is a common symptom in patients with atopic dermatitis and psoriasis. Patients with atopic dermatitis and psoriasis often report pruritis-associated sleep impairments and scratching behaviors during nighttime and the negative impact on their quality of life. However, nocturnal scratch behavior and sleep impairment are poorly understood due to the difficulties in quantifying these symptoms in patients' daily lives. This study deploys multiple technologies (polysomnography, video capture, wrist sensors, clinician-reported outcomes, and patient-reported outcomes) to develop and validate a wrist-based solution to quantify nocturnal scratch.

ELIGIBILITY:
Inclusion criteria for participants with atopic dermatitis:

* At least 14 years old
* Less than 70 years old
* Clinical diagnosis of Atopic Dermatitis
* Peak Pruritis NRS score > 1

Inclusion criteria for participants with psoriasis:

* At least 18 years old
* Less than 70 years old
* Clinical diagnosis of plaque psoriasis
* At least a peak pruritis PNRS of 4
* Itch is caused by psoriasis, as determined by clinician

Exclusion Criteria:

* Non-Atopic Dermatitis or Psoriasis-related sleep disorder (e.g., diagnosed sleep apnea, restless leg syndrome etc...)
* Movement disorder
* Flare or infection on the wrist
* Infected atopic dermatitis or psoriasis lesions
* Pregnant or lactating women
* Shift workers or participants with jetlag
* Current diagnosis of depression

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female subjects, aged 14-70 years old, with active atopic dermatitis or psoriasis
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Scratch Movements | 14 days
  To evaluate the agreement in the detection of scratching behaviour between video annotation and wrist-based sensor
Sleep Time | 14 days
  To evaluate the agreement in the detection of sleep patterns between polysomnography and wrist-based sensor

CONTACTS AND LOCATIONS:
Overall Officials: Damien Leger, Principal Investigator — Université Paris Cité, VIFASOM, ERC 7330, Paris, France;b AP-HP, Hôtel-Dieu, Centre du Sommeil et de la Vigilance, Paris, France
Locations (1):
- AP-HP, Hôtel-Dieu, Centre du Sommeil et de la Vigilance, Paris, France